CLINICAL TRIAL: NCT03618433
Title: KİNECT® - Video Games Based Physiotherapy Programme in Patients With Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özlem Feyzioğlu, MSc, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATADEK-2018 / 9
Record Dates: First submitted 2018-07-30; First posted 2018-08-07 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Upper Extremity Dysfunction; Mastectomy
Keywords: kinect; breast cancer; mastectomy; upper extremity dysfunction
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Standart exercise protocol and KİNECT® video based physiotherapy
  The treatment protocol of the study group will consist of soft tissue massage, passive mobilization, stretching, self-stretching exercises.In total, a 25-minute Kincet® video game program will be applied in addition to the 15-minute basic and standart exercise program.
  Interventions: Other: study group
- Control group (Active Comparator): Standart exercise protocol and Upper extremity rehabilitation
  The control group included soft tissue massage, stretching, self-stretching, passive mobilization, coordination, posture exercises, progressive active and assisted shoulder exercises, proprioception and strengthening exercises in the exercise therapy protocol
  Interventions: Other: Control group

INTERVENTIONS:
Other: study group — The treatment protocol will consist of soft tissue massage, passive mobilization, stretching, self-stretching exercises. and shoulder proprioception .In addition to the standart exercise therapy, Kincet® video game program will be applied .
  Other Names: Kinect based therapy and standart exercise
  Arms: Study group
Other: Control group — The control group included soft tissue massage, stretching, self-stretching, passive mobilization, coordination, posture exercises, progressive active and assisted shoulder exercises, proprioception and strengthening exercises in the exercise therapy protocol
  Other Names: Standart exercise and upper extremity rehabilitation
  Arms: Control group

SUMMARY:
The main objective of the study is to investigate the effects of Kinect® video based technology on pain, functionality, muscle strength, fatigue and quality of life in patients with breast cancer surgery and axillary node dissection.

DETAILED DESCRIPTION:
Introduction: Breast cancer is the most common cancer seen in women. 1.7 million new cases have been reported in the world and have been shown as the fifth cause of death among women.There are many risk factors in etiogenesis, including gender, family history, age, obesity, malnutrition in postmenopausal period, hormone therapy, after 30 years of first birth, alcohol consumption and physical activity inadequacy. Pain and functional disorders are common complications after post-mastectomy in upper extremity. After mastectomy surgery ,pain in the shoulder, fatigue, decrease in range of motion, restriction of daily living activities, decrease of muscle strength, postural inbalance,, neuropathy and lymphedema may occur in the acute and chronic period.

Patients with breast cancer need a multidisciplinary and ongoing physiotherapy program.New technologies provide more motivational involvement for patients according to regular care and standard programs. Microsoft Kinect® is a virtual exercise program that is an application. It has been in use for rehabilitation among physical therapists for different deseas.The Kinect® application is a special technological approach that allows to follow the movements of the body. Microsoft Kinect® virtuel reality video games are promissing rehabilitation options because they involve upper extremity practise.

Subjects and methods: A randomized clinical trial, the examiner being blinded unaware of the intervention group to which subjects were assigned. Participants will be randomly assigned to two groups:

Experimental group- where the participants will be treated with standart exercise therapy and Kinect® video-game-based technology

Control Group - Standart exercise therapy and upper extremity rehabilitation-oriented physiotherapy program will be applied.

The evaluations will be repeated at the beginning of the study and at the end of the sixth week. Data obtained from the study will be analyzed using appropriate statistical methods. Patients will be received to therapy which upper extremity rehabilitation or Kinect based video game play under physiotherapist supervision for two days a week for six weeks. Patients will be supported by the home exercise program, except during sessions. Participants' joint range of motion in the initial assessments will be measured by electro-goniometer, muscle strength assessment by JTech hand dynamometer at appropriate evaluation positions and grip force asssessment by Saehan Hydraulic Hand Dynamometer . In assessing pain, pain levels at rest and during activity will be questioned using Visual Analog Scale. Fear of movement of individuals will be assessed via Tampa Kinesiophobia Scale and functional levels will be assessed via Disabilities of the Arm Shoulder and Hand Anketi (DASH). Environmental measurement differences between upper extremities with and without operation will be assessed with made in the arm, forearm and the wrist. In assessing Quality of life will be assessed European Organization for Research and Treatment of Cancer EORTC QLQ-C30 - EORTC- BR23 and finally fatique of individuals will be assessed via Cancer Fatigue Scale -CFS.

Sample size: 17 women for each group. Data Analysis:Data obtained from the study will be analyzed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer and having axillary lymph node dissection,
* Post -operative in two weeks,
* VAS score>1,
* Women who do not present contraindications for physiotherapy (infection, metastasis, locoregional recurrence)
* Women who have read, understood and signed informed consent freely

Exclusion Criteria:

* Patients who had breast cancer surgery contralateral or the same side before
* active or metastatic cancer centers
* a neurological condition or orthopedic surgery that affects upper extremity function
* pacemaker, infection, open wound,
* Women with cognitive limitations to understand the information provided, instructions for treatment and consent to their participation in the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Range of motion | 6 weeks
  Shoulder range of motion will be evaluated by digital goniometer. Shoulder flexion degree, shoulder extension degree, abduction and adduction degree, internal rotation and external rotation degree will be assessed with digital goniometer. The results will be recorded in degrees.

SECONDARY OUTCOMES:
Pain - Visual Analogue Scale- | 6 weeks
  Visual Analogue Scale is one of the simple and common methods used in pain assessment. Self reported pain intensity during the rest and the activity measured by 0-10 centimeter chart. Visual Analogue Scale (VAS), where 0 indicates no pain or best and 10 indicates the most intense pain imaginable or worst. The patient will mark the severity of the pain on a 10 cm long chart.
Muscle strength | 6 weeks
  Hand-held dynamometer will be used to evaluate shoulder muscles' strength
Circumference | 6 weeks
  Upper arm circumference (millimeters) was measured to the nearest millimeter with a steel tape. Measurement will be made wrist, with 10 cm proximal of the wrist, at the lateral epicondyle, and 10 cm proximal of the elbow while arm hanging relaxed.
Grip strength | 6 weeks
  Grip strength was evaluated by hand grip dynamometry (Saehan Hydraulic Hand Dynamometer ) Measurements were performed in affected side according to positions defined by American Society of Hand Therapists (sitting with the shoulder adducted to the side and the elbow flexed 90° with the forearm and wrist in the neutral mid-position)
Fatigue | 6 weeks
  The Cancer Fatique scale (CFS) will be used to evaluate fatique. The cancer fatigue scale (CFS) was developed for the purpose of identifying and measuring fatigue in cancer patients, and its validity was evaluated in cancer patients and also in a scale determined specifically in breast cancer cases.The scale consists of 15 items and three subscales; physical, affective, and cognitive. Each item is scored between 1 and 5. 1 is never asked, 5 is too much.The high score indicates the excess of fatigue severity.The maximum total score is 60.

OTHER OUTCOMES:
Disabilitiy | 6 weeks
  Disabilities of the Arm Shoulder and Hand ( DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms.The DASH questionnaire consists of three parts.The first part consists of 30 questions. 21 questions assess the difficulty of the patient in daily life activities, 5 question symptoms, and the remaining 4 questions assess social function, work, sleep, and self-confidence of the patient.In the DASH questionnaire, questions are answered in 5-point likert system. 1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not at all. The total score varies between 0 and 100 points and the low score indicates good health.
Kinesiophobia | 6 weeks
  Tampa Kinesiophobia Scale will be used to assess the fear of movement. It is a 17-item self report checklist using a 4-point Likert scale that was developed as a measure of fear of movement or (re)injury. 1 = Absolutely not, 4 = Completely agree.When the total score is between 17 and 68, a higher score means that there is more fear of movement.
Qualitiy of Life - European Organization for Research and Treatment of Cancer EORTC QLQ-C30 - EORTC- BR23 | 6 weeks
  The European Organization for Research and Treatment of Cancer EORTC QLQ-C30 (version 3.0) is a cancer-specific measure of life quality. It consists of 30 items to assess physical, role, emotional, cognitive and social functioning, global health status or qualitiy of life scales, fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties. The EORTC QLQ-BR23 is a breast-specific module that comprises of 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss.All scores will linearly transforme to a 0 to 100 scale. A high or healthy level of functioning is represented by a high functional score. More severe symptoms or problems are represented by high symptom scores or items.

CONTACTS AND LOCATIONS:
Locations (1):
- Okemeydanı Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feyzioglu O, Dincer S, Akan A, Algun ZC. Is Xbox 360 Kinect-based virtual reality training as effective as standard physiotherapy in patients undergoing breast cancer surgery? Support Care Cancer. 2020 Sep;28(9):4295-4303. doi: 10.1007/s00520-019-05287-x. Epub 2020 Jan 6. PMID 31907649